CLINICAL TRIAL: NCT00922909
Title: Executive Control Analysis in Patients Suffering From Parkinson Disease and Treated by Deep Brain Stimulation (Chronometric and Electromyographic Approach During a Simon Task)
Brief Title: Executive Control Analysis in Patients Suffering From Parkinson Disease and Treated by Deep Brain Stimulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 2009/14; 2009-A00333-54
Record Dates: First submitted 2009-06-16; First posted 2009-06-17 (Estimated); Last update posted 2014-02-25 (Estimated); Status verified 2014-02

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- 2 (Active Comparator): Day 1 : morning : Medication on ; Stimulation : off afternoon : Medication : on ; Stimulation : on Day 2 : morning : Medication : off ; Stimulation : off afternoon : medication : off ; stimulation : on
  Interventions: Behavioral: Simon task
- 3 (Active Comparator): Day 1 : morning : Medication off ; Stimulation : on afternoon : Medication : off ; Stimulation : off Day 2 : morning : Medication : on ; Stimulation : on afternoon : medication : on ; stimulation : off
  Interventions: Behavioral: Simon task
- 4 (Active Comparator): Day 1 : morning : Medication off ; Stimulation : off afternoon : Medication : off ; Stimulation : on Day 2 : morning : Medication : on ; Stimulation : off afternoon : medication : on ; stimulation : on
  Interventions: Behavioral: Simon task
- 1 (Active Comparator): Day 1 : morning : Medication on ; Stimulation on afternoon : Medication on ; Stimulation off Day 2 : morning : Medication off ; Stimulation on afternoon : Medication off ; Stimulation off
  Interventions: Behavioral: Simon task

INTERVENTIONS:
Behavioral: Simon task — Reaction time task

SUMMARY:
Different results have recently led to question the classical notion according to which the motor and cognitive deficits in Parkinson's disease are tied to a thalamo-cortical inhibition due to the degeneration of the dopaminergic nigro-striatal pathways. Instead, Parkinsons's disease seems accompanied by an increase in motor cortical activity.

A reaction time task, known as the "Simon task" in the literature, allows one to study the influence of irrelevant visual information on decision making. In the most common version of this task (used in the prosed study), the subjects have to choose between a left- and a right-hand keypress according to the color of a visual signal presented either to the left or to the right of a fixation. The to be established association is said "congruent" when the response is ipsilateral to the stimulus and "incongruent" when the response is contralateral to the stimulus. In healthy volunteers, EMG investigations have revealed that in a significant numbers of trials, the contraction of the response agonist is preceded by a infra-liminal contraction of the agonist involved in the non-required response. Such "partial errors" demonstrate that the nervous system is able to detect, abort and correct a part of its errors, thereby revealing the existence of an on-line executive control in simple decision tasks. Behavioral studies performed in Parkinson disease patients, suggest that these patients may experience a deficit in such a control.

The present study aims at testing this hypothesis by assessing the effect of subthalamic stimulation on the patients' performance in a Simon task.

DETAILED DESCRIPTION:
Different results have recently led to question the classical notion according to which the motor and cognitive deficits in Parkinson's disease are tied to a thalamo-cortical inhibition due to the degeneration of the dopaminergic nigro-striatal pathways. Instead, Parkinsons's disease seems accompanied by an increase in motor cortical activity.

A reaction time task, known as the "Simon task" in the literature, allows one to study the influence of irrelevant visual information on decision making. In the most common version of this task (used in the prosed study), the subjects have to choose between a left- and a right-hand keypress according to the color of a visual signal presented either to the left or to the right of a fixation. The to be established association is said "congruent" when the response is ipsilateral to the stimulus and "incongruent" when the response is contralateral to the stimulus. In healthy volunteers, EMG investigations have revealed that in a significant numbers of trials, the contraction of the response agonist is preceded by a infra-liminal contraction of the agonist involved in the non-required response. Such "partial errors" demonstrate that the nervous system is able to detect, abort and correct a part of its errors, thereby revealing the existence of an on-line executive control in simple decision tasks. Behavioral studies performed in Parkinson disease patients, suggest that these patients may experience a deficit in such a control.

Aims

The present study aims at testing this hypothesis by assessing the effect of subthalamic stimulation on the patients' performance in a Simon task.

Methods

Sixteen non-demented Parkinson disease patients treated by deep brain stimulation will be involved in the study. They will perform a Simon task in four conditions: Stimulator ON vs. OFF x Medication ON vs. OFF. The EMG activity of the response agonist will be recorded during task performance. Such recordings will allow the investigator to uncover partial errors. This index together with reaction time and overt errors will be subsequently analysed.

Expected results

Deep brain stimulation (as oral Dopaminergic medication) re-install the patient motor functions and it is thus predicted that both the stimulation and the medication improve the patients executive control by increasing the proportion of partial errors relative to overt errors. Such a result would demonstrate that the nigro-striatal pathways in directly involved in executive control during decision making.

ELIGIBILITY:
Inclusion Criteria:

* Parkinson disease
* Mattis score > 130,MMSE > 24
* No subthalamic stimulation for 6 months
* No depressive disease evoluting

Exclusion Criteria:

* Colorblindness
* Psychotropic treatment introduced for less than a month

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2009-06; Primary Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
to assess the effect of subthalamic stimulation on the patients' performance in a Simon task. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Philippe AZULAY, Principal Investigator — Assistance Publique-Hôpitaux de Marseille
Locations (1):
- Assistance Publique-Hopitaux de Marseille, Marseille, France